CLINICAL TRIAL: NCT06007443
Title: Association Between Pain Related Variables in Patients With Chronic Neck Pain
Brief Title: Pain Related Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Kübra Canli, Principal investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CPM-TS-2PD
Record Dates: First submitted 2023-07-04; First posted 2023-08-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-08

CONDITIONS: Chronic Neck Pain; Musculoskeletal Pain; Pain Modulation; Cortical Plasticity; Conditioned Pain Modulation; Temporal Summation
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with neck pain (Experimental): conditioned pain modulation, temporal summation and two-point discrimination will be evaluated in all included participants. Average pain intensity will be asked
  Interventions: Other: pain related variables assessment

INTERVENTIONS:
Other: pain related variables assessment — Pressure pain threshold, conditioned pain modulation, temporal summation, and two-point discrimination will be evaluated on the upper trapezius muscle. Average pain intensity will be asked.

SUMMARY:
Chronic neck pain is a common problem among the general population. Patients with chronic neck pain used health care services twice as much as the population on average, mainly due to intense pain intensity. It is well-known that pain intensity depends on the association of pain processing in several levels of central pain processing.

Identifying the association between conditioned pain modulation, temporal summation, and somatosensory representation, all represent separate central pain processing, will provide an opportunity to develop treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* pain in the back of the neck region
* pain longer than 3 months
* pain intensity at least 3 based on the visual analog scale

Exclusion Criteria:

* vertebra fracture
* fibromyalgia
* chronic fatigue syndrome
* surgery to the neck or shoulder
* radicular pain
* neurologic deficit due to disk hernia
* spinal stenosis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-01-28 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
pressure pain threshold | 'baseline'
  The pressure pain threshold (PPTs) of the upper trapezius and dominant tibialis anterior muscles will be evaluated. For the upper trapezius muscle, assessment will be made approximately 5 to 8 cm superomedial to the superior angle of the scapula. For the tibialis anterior muscle, the assessment will be made muscle belly, which is approximately 2.5 cm lateral and 5 cm inferior to the tibial tubercle. Palpation during resisted active dorsiflexion ensured that the tibialis anterior muscle belly had been found.
  Pressure pain thresholds will assessed using a pressure algometer (Algometer) with a stimulation area of 1 cm2. The increment rate of pressure will be kept at approximately 1 kg/cm2/s. The first time the pressure perceived as pain will be recorded as a PPTs. Two PPT assessments with a 30 second will be completed, and the average was used for statistical analysis.

SECONDARY OUTCOMES:
temporal summation | 'baseline'
  Temporal summation (TS) of pressure pain will be elicited at the upper trapezius muscle by administering 10 consecutive pressure pulses using the algometer. For each pulse of the TS procedure, the pressure will be increased at approximately 2 kg/s until the previously determined PPT will be reached and maintained for one second. Pressure pulses will be presented with an inter-stimulus interval of one second. Participants will be instructed to rate their perceived pain intensity during the first, fifth, and tenth pressure pulse using a verbal numeric rating scale (VNRS). The TS pain score will be obtained by subtracting the first VNRS score from the last VNRS, with increased number indicates higher pain facilitation
conditioned pain modulation | 'baseline'
  An inflated occlusion cuff placed on the contralateral arm will be used as a conditioned stimulus. The occlusion cuff will be inflated at a rate of 20 mm Hg/s until "the first sensation of pain". At that point, it will be maintained for 30 s. Pain intensity will then be rated on a VNRS. Next, cuff inflation will be increased or decreased until the VNRS will be rated as 3/10. PPTs assessment will be repeated during maintenance of the cuff inflation. CPM will be calculated as the first NRS score during cuff inflation minus the first VNRS score before cuff inflation, with more positive values indicating more pain inhibition and more negative values indicating more pain facilitation.
tactile acuity | 'baseline'
  It will be assessed by using two-point discrimination threshold on both sides of the neck.
  A sliding two-point Vernier Calliper with digital measurement will be placed under its own weight on the participant's skin, to provide two simultaneous tactile stimuli. For the spinal measures, the caliper will be aligned vertically 15 mm lateral to the spinous processes of C7. Assessment will be commenced with the two-points at a 20 mm separation, and will be increased by 2 mm increments until the participant reported feeling two points of contact. If two distinct points perceived in three consecutive trials this value will be recorded. A series of three ascending and descending assessments will be performed, with the mean of the six values will be used for analyses.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)